CLINICAL TRIAL: NCT03078985
Title: Cardiovascular Magnetic Resonance-Guided Radiofrequency-Ablation for Atrial Flutter
Brief Title: Cardiovascular Magnetic Resonance-Guided Radiofrequency-Ablation for Atrial Flutter II
Acronym: 2016-IMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other); Philips Healthcare (Industry); Imricor Medical System (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-IMR
Record Dates: First submitted 2016-12-10; First posted 2017-03-14 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Atrial Flutter
Keywords: real-time MRI; electrophysiology study; atrial flutter ablation; active tracking
MeSH Terms: conditions — Atrial Flutter | interventions — Catheter Ablation

STUDY DESIGN:
Masking Description: This an Open Label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ablation for typical atrial flutter (Experimental): This group receives an MR-guide ablation for atrial flutter with the study device ( Vision-MR ablation catheter )
  Interventions: Procedure: ablation for typical atrial flutter; Device: catheter ablation with study device

INTERVENTIONS:
Procedure: ablation for typical atrial flutter — Typical atrial flutter is treated by catheter ablation.
Device: catheter ablation with study device — The study device is used inside the MRI environment to localize the cavotricuspid isthmus (CTI). The CTI is then treated with radiofrequency energy to achieve complete isthmus block.

SUMMARY:
The purpose of this clinical study is to assess the safety and performance of the Vision-MR Ablation Catheter, the primary safety endpoint will measure the rate of serious adverse events related to the device or procedure; the primary performance endpoint will measure the acute success rate defined as the demonstration of bidirectional cavo-tricuspid isthmus block after radiofrequency application in the cavo-tricuspid isthmus; the secondary performance endpoint will measure the chronic success rate defined as the freedom of recurrence of type 1 atrial flutter at three months post-ablation procedure. The study will be a single center study conducted at the Leipzig University Hospital Heart Center in Germany. The study population will consist of adult patients requiring ablation for type I atrial flutter.

This is the follow-up study to NCT02699034.

DETAILED DESCRIPTION:
The study will be a single center study conducted at the Leipzig University Hospital Heart Center in Germany. 35 subjects subjects meeting inclusion/exclusion criteria will participate in the study. This study requires the use of investigational products from two independent manufacturers: Imricor and Philips. Imricor has developed the ablation catheter with related accessory cables and electrophysiology (EP) recorder/stimulator system. Philips has developed an image guidance and mapping system that is compatible with the Imricor products.

The Vision-MR Ablation Catheter will be used in conjunction with the following investigational products: Vision-MR Ablation Cable Set, Vision-MR Diagnostic Cable, the interventional MRI Suite (iSuite) image guidance and mapping system, and a dStream Interface (dSIF-FE). With the exception of iSuite and dSIF-FE, which are manufactured by Philips, Imricor will provide all investigational devices used in the study.

Each procedure will require two single-use Vision-MR Ablation Catheters and one each of the two single-use accessory catheter cables.

Ablation for the treatment of arrhythmia is an inherently complex procedure. Use of the investigational products listed above under MR guidance is an emerging approach to performing the interventional electrophysiology procedure.

The study population will consist of adult patients requiring ablation for type I atrial flutter.

Study subjects will require a follow-up visit or telephone call at seven days post procedure. Accordingly, the expected total study duration is approximately 9 months with study start planned for February 2017.

This is the follow-up study to NCT02699034 which was terminated early based on a recommendation by the oversight authority. The study device (Vision-MR ablation catheter) has been improved and the EP recorder/stimulator is now CE-marked.

ELIGIBILITY:
Inclusion Criteria:

* First time indication for ablation for type I atrial flutter.
* Patients willing and able (mentally and physically capable per physician's discretion) to understand the investigational nature, potential risks and benefits of the study and able to provide written informed consent to participate in the study and agree to comply with follow-up visits and evaluation
* Patients able to receive anticoagulation therapy to achieve adequate anticoagulation

Exclusion Criteria:

* Contraindication for MRI diagnostic exam
* A cardiac ablation or cardiac surgery within 180 days prior to enrollment
* Documented intracardiac thrombus, tumor, bleeding, clotting or other abnormality that precludes catheter introduction and placement
* Myocardial infarction within 60 days prior to enrollment
* Current unstable angina
* History of cerebrovascular event (within 180 days prior to enrollment)
* Patients with an ejection fraction less than or equal to 35% within 90 day prior to enrollment
* Permanent leads in or through the right atrium
* Clinically significant structural heart disease (including tricuspid valve regurgitation, tricuspid valve stenosis or other congenital heart disease) that would preclude catheter introduction and placement, as determined by the Investigator
* Uncompensated congestive heart failure (NYHA Class III or IV)
* Arrhythmia is secondary to electrolyte imbalance, thyroid disease, or other reversible or non-cardiovascular cause
* Known sensitivity to heparin or warfarin
* Active or systemic infection
* Any other significant uncontrolled or unstable medical condition (including but not limited to hypertension and diabetes)
* contraindication for conventional ablation procedure know allergy against radiocontrast agents renal insufficiency with glomerular filtration rate < 30ml/min/1,73m2
* Women who are pregnant or plan to become pregnant within the course of their participation in the investigation or who are breastfeeding
* Life expectancy of less than 12 months
* Patients with prosthetic valves
* Contraindicated for transfemoral venous access
* Older than 75 years
* Current enrollment in any other clinical investigation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with bidirectional cavo-tricuspid isthmus block after intervention | 9 months
  Acute success defined as the demonstration of the established electrophysiological endpoint (e.g. bidirectional cavo-tricuspid isthmus block after radiofrequency application in the cavo-tricuspid isthmus) with the investigational device. Historically, the acute success rate for RF ablation of type I atrial flutter is 85%. Analysis will be based on a binomial proportion and expressed as a percentage. For a total of N subjects with S achieving success, the percentage, represented as P, will be calculated as P = 100*S/N.
Number of patients with periinterventional serious adverse events | 9 months
  The primary safety endpoint is the rate of serious adverse events (SAEs) related to the device or procedure assessed at the 7-day follow-up. Analysis will be based on a binomial proportion and expressed as a percentage. For a total of N subjects with S experiencing an SAE related to the device or procedure, the percentage, represented as P, will be calculated as P = 100*S/N.
Number of patients with freedom from recurrence from type I atrial flutter 3 months (chronic success rate) after ablation (study procedure). | 9 month
  The primary chronic performance endpoint is the chronic success rate defined as freedom from recurrence of type 1 atrial flutter at 3 months post procedure. Freedom of recurrence of type I atrial flutter is assessed using symptom survey, ECG and echocardiogram data. This will be evaluated separately for all subjects treated with the device and for all subjects that achieved acute success (defined by the primary acute performance endpoint).

SECONDARY OUTCOMES:
Number of patients with freedom from recurrence from type I atrial flutter 6 months after ablation (study procedure). | 9 month
  The secondary performance endpoint is the chronic success rate defined as freedom from recurrence of type 1 atrial flutter at 6 months post procedure. Freedom of recurrence of type I atrial flutter is assessed using symptom survey, ECG and echocardiogram data. This will be evaluated separately for all subjects treated with the device and for all subjects that achieved chronic success (defined by the primary chronic acute performance endpoint).

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Center Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hilbert S, Sommer P, Gutberlet M, Gaspar T, Foldyna B, Piorkowski C, Weiss S, Lloyd T, Schnackenburg B, Krueger S, Fleiter C, Paetsch I, Jahnke C, Hindricks G, Grothoff M. Real-time magnetic resonance-guided ablation of typical right atrial flutter using a combination of active catheter tracking and passive catheter visualization in man: initial results from a consecutive patient series. Europace. 2016 Apr;18(4):572-7. doi: 10.1093/europace/euv249. Epub 2015 Aug 27. PMID 26316146
- [Background] Grothoff M, Gutberlet M, Hindricks G, Fleiter C, Schnackenburg B, Weiss S, Krueger S, Piorkowski C, Gaspar T, Wedan S, Lloyd T, Sommer P, Hilbert S. Magnetic resonance imaging guided transatrial electrophysiological studies in swine using active catheter tracking - experience with 14 cases. Eur Radiol. 2017 May;27(5):1954-1962. doi: 10.1007/s00330-016-4560-7. Epub 2016 Aug 23. PMID 27553931
- See also: Imricor website — http://www.imricor.com